CLINICAL TRIAL: NCT07070999
Title: A Phase 1-2, Open-Label, Multicenter Study to Assess the Safety, Tolerability and Efficacy of a Single Dose of GB221 Delivered Into the Cisterna Magna of Pediatric Participants From 2 Weeks to Younger Than 12 Months of Age With Spinal Muscular Atrophy Type 1
Brief Title: Study of Safety, Tolerability and Efficacy of GB221 in Infants With Spinal Muscular Atrophy Type 1
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gemma Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GB221-101; CHARISMA (Other: Gemma Bio, Inc.)
Record Dates: First submitted 2025-05-30; First posted 2025-07-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Spinal Muscular Atrophy Type I
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1A, safety and exploratory efficacy of a single dose in symptomatic participants (Experimental): Symptomatic participants with SMA Type 1 (up to 3 copies of SMN2), who are either treatment naïve or receiving risdiplam, with onset of disease during the first 6 months of life, aged from 2 weeks to younger than 12 months at the time of dosing.
  Interventions: Biological: GB221
- Cohort 1B, expansion phase for confirmatory testing in symptomatic participants (Experimental): Symptomatic participants with SMA Type 1 (up to 3 copies of SMN2), who are either treatment naïve or receiving risdiplam, with onset of disease during the first 6 months of life, aged from 2 weeks to younger than 12 months at the time of dosing.
  Interventions: Biological: GB221
- Cohort 2A, safety and exploratory efficacy of a single dose in presymptomatic participants (Experimental): Presymptomatic participants (treatment naïve or receiving risdiplam) at risk of developing SMA Type 1 (up to 2 copies of SMN2), aged from 2 weeks to younger than 5 months (< 150 days) at the time of dosing.
  Interventions: Biological: GB221
- Cohort 2B, expansion phase for confirmatory testing in presymptomatic participants (Experimental): Presymptomatic participants (treatment naïve or receiving risdiplam) at risk of developing SMA Type 1 (up to 2 copies of SMN2), aged from 2 weeks to younger than 5 months (< 150 days) at the time of dosing.
  Interventions: Biological: GB221

INTERVENTIONS:
Biological: GB221 — GB221

SUMMARY:
GB221 is a gene therapy that delivers a working SMN1 gene to the motor neurons of people with spinal muscular atrophy (SMA) Type 1. This study will evaluate the safety, tolerability and efficacy of GB221 in two groups:

1. participants aged from 2 weeks to younger than 12 months presenting with symptoms of SMA Type 1 who have never received a treatment OR are receiving the drug risdiplam
2. participants aged from 2 weeks to younger than 5 months who are at risk of developing SMA Type 1 (presymptomatic) and have never received treatment OR are receiving the drug risdiplam.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Participants

  1. Diagnosis of SMA Type 1 based on gene mutation analysis with bi-allelic SMN1 mutations (deletion or point mutations) and up to 3 copies of SMN2
  2. Participants must be 2 weeks to < 12 months of age at the time of dosing with disease onset of during the first 6 months of life.
* Presymptomatic Participants

  1. At risk of SMA Type 1 based on gene mutation analysis with bi-allelic SMN1 mutations (deletion or point mutations) and up to 2 copies of SMN2
  2. Participants must be 2 weeks to < 5 months (< 150 days) of age at the time of dosing.

Exclusion Criteria:

1. Any suspected or confirmed active viral infection at screening baseline (including HIV, Hepatitis B or C, or human T Cell lymphotropic viruses [HTLV])
2. History of invasive ventilatory support (tracheotomy with positive pressure) or pulse oximetry <95% saturation.
3. Ongoing immunosuppressive therapy or immunosuppressive therapy within 3 months of starting the trial (e.g. corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab)
4. Participation in a recent SMA treatment clinical trial that, in the opinion of the Investigator, creates unnecessary risks for gene transfer.
5. Prior history of gene therapy for any indication, hematopoietic transplant or solid organ transplant
6. Subjects with severe scoliosis
7. Known allergy or hypersensitivity to prednisolone or other glucocorticosteroids or their excipients.

Ages: 2 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (AEs) and serious adverse events (SAEs) at Grade 3 or higher as characterized by CTCAEv5.0 | Up to 18 months across multiple visits
  Assess the number of treatment-related AEs and SAEs as characterized by CTCAEv5.0
Number of Participants with Clinically Significant Changes in Physical Functions | Up to 18 months across multiple visits
  Assess the number of participants with clinically significant changes in physical functions.
Number of Participants with Clinically Significant Changes in Neurological Functions | Up to 18 months across multiple visits
  Assess the number of participants with clinically significant changes in neurological functions.
Number of Participants with Clinically Significant Changes in Vital signs | Up to 18 months across multiple visits
  Assess the number of participants with clinically significant changes in vital signs.
Change in electrocardiogram results | Up to 18 months across multiple visits
  ECG will measure RR interval, P Wave, PR interval, PR segment, QRS Complex, ST segment, T wave and QT Interval.
Change in serum cardiac troponin I levels | Up to 18 months across multiple visits
Number of Participants with Clinically Significant Laboratory Abnormalities as Measured Using Hematology, Chemistry and Coagulation Tests | Up to 18 months across multiple visits
  Assess the number of participants with clinically significant laboratory changes including hematology, serum chemistry, and coagulation tests.
Number of Participants with Clinically Significant Laboratory Abnormalities as Measured Using Urine and CSF Tests | Up to 18 months across multiple visits
  Assess the number of participants with clinically significant laboratory changes including urine and CSF tests.
Change in markers of immunogenicity | Up to 18 months across multiple visits
  Assessment of humoral (NAb and TAb titers) and T-cell (IFNγ ELISpot) immune responses to the AAVhu68 capsid and SMN transgene product in serum and CSF.

SECONDARY OUTCOMES:
Assess the number of participants who experience permanent ventilation or death | Up to 18 months across multiple visits
Percentage of infants with improvement in the motor milestones categories in Section 2 of the Hammersmith Infant Neurological Examination (HINE), with the exclusion of voluntary grasp. | Baseline, 6 months and 18 months post dose.
  * improvement in at least one category, i.e., an increase in the score for head control, rolling, sitting, crawling, standing, or walking of ≥1 point,
  * an increase in the score for kicking of ≥2 points, or achievement of the maximal score for kicking.
Change from baseline in mean Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) Score. | Baseline, 6 months and 18 months post dose.
  Assess 16 types of muscle movements, each given a score from zero (the person can't complete the movement) to 4 (the person can complete the movement on their own, without assistance) to produce a score of 0 to 64.

CONTACTS AND LOCATIONS:
Overall Officials: May Orfali, MD, Study Director — Gemma Biotherapeutics

IPD SHARING:
Plan to Share IPD: No